CLINICAL TRIAL: NCT01492348
Title: Stepped Enhancement of PTSD Services Using Primary Care (STEPS UP): A Randomized Effectiveness Trial
Acronym: STEPS UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); RAND (Other); RTI International (Other); University of Washington (Other); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-09-2-0077
Record Dates: First submitted 2010-03-31; First posted 2011-12-14 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Depression
Keywords: collaborative care; PTSD; military; Depression; primary care; care management; stepped care; telehealth; OIF; OEF; preference-based treatment; cost effectiveness; web-based treatment; telephonic CBT; evidence-based treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPS UP Intervention (Experimental): STEPS UP is a centrally assisted stepped collaborative telecare management program within primary care. The STEPS UP intervention added to Optimized Usual Care (PCMH-BH; formerly RESPECT-Mil) in 4 ways: (1) care management enhancements; (2) stepped psychosocial treatment options (web, phone, in person); (3) electronic symptom registry for measurement-based treatment planning (symptoms are measured at regular intervals and care is intensified for patients with recurrent or persistent PTSD and/or depressive) and for telecare manager caseload and site performance monitoring; and (4) routine assisted review of patient, telecare manager, and site performance by a central psychiatrist and psychologist.
  Interventions: Behavioral: STEPS UP
- Optimized Usual Care (OUC) (Active Comparator): Service members randomized to Optimized Usual Care (OUC) will get usual treatment at the site. OUC is RESPECT-Mil, a voluntary, primary care-based implementation program where, with the assistance and collaboration of a psychiatrist and an on-site nurse-level care manager, service members with symptoms of PTSD and depression are screened, tracked, and treated within the primary care system.
  Interventions: Behavioral: OUC

INTERVENTIONS:
Behavioral: STEPS UP — The STEPS UP intervention enhances RESPECT-Mil in several ways:
  1. Adds care manager training in motivational enhancement, problem solving, and behavioral activation strategies to improve patient engagement.
  2. Adds preference-based stepped care (i.e., order of steps determined by symptom severity, patient preference, & primary care recommendation) to existing options of pharmacotherapy that includes web-based self-management programs; flexible, modularized telephone-delivered CBT; and individual face to face psychotherapy by specialist.
  3. Adds option for centralized, telephone-based care management to improve fidelity of intervention delivery, continuity of care, and access to care during off-hours.
  4. Adds a centralized care team using an electronic symptom registry to provide staffing to care managers, track patients longitudinally, develop stepped-based treatment recommendations, and monitor intervention components.
  Arms: STEPS UP Intervention
Behavioral: OUC — Service members randomized to Optimized Usual Care (OUC) will get usual treatment at the site. OUC is RESPECT-Mil, a voluntary, primary care-based implementation program based on the "three-component model" where, with the assistance and collaboration of a psychiatrist and an on-site nurse-level care manager, service members with symptoms of PTSD and depression are screened, tracked, and treated within the primary care system. Components of the RESPECT-Mil program include (1) equipping and training primary care clinics to screen each visit and use symptom severity tools for diagnosis and assessment; (2) using nurse care managers to assist patients and primary care clinicians; and (3) increasing access to a mental health specialist, often using a clinic specialist.
  Arms: Optimized Usual Care (OUC)

SUMMARY:
The overall objective of this study is to test the effectiveness of a systems-level approach to primary care recognition and management of PTSD and depression in the military health system. More specifically, the investigators will test the effectiveness of a telephone care management with preference-based stepped PTSD/depression care--STepped Enhancement of PTSD Services Using Primary Care (STEPS UP)--as compared to Optimized Usual Care (OUC).

Primary Hypothesis 1: Active duty primary care patients with PTSD, depression, or both who are randomly assigned to STEPS UP will report significantly greater reductions in PTSD and depression symptom severity compared to participants assigned to OUC over 12-months of follow-up.

Hypothesis 2: Active duty primary care patients with either PTSD, depression, or both who are randomly assigned to STEPS UP will report significantly greater improvements in somatic symptom severity, alcohol use, mental health functioning, and work functioning compared to participants assigned to OUC over 12-months of follow-up.

Hypothesis 3: The STEPS UP program will be both more costly and more effective compared to OUC over the 12-months of follow-up, and will have a favorable cost-effectiveness ratio in terms of dollars per quality adjusted life years saved.

Hypothesis 4: Active duty primary care patients participating in STEPS UP, their clinicians, care managers, and family members will report that STEPS UP is acceptable, effective, satisfying, and appropriate PTSD and depression care.

DETAILED DESCRIPTION:
Despite the significant prevalence of posttraumatic stress disorder (PTSD) and depression among veterans returning from Operations in Iraq and Afghanistan, less than half of service members who are referred for a specialty mental health assessment actually receive specialty mental health treatment. Systematic knowledge regarding access to care and quality of care delivered in civilian, VA, and military facilities for those who encounter barriers or difficulty is scant, and recent policy reviews have strongly questioned availability and quality of care. These problems of access and quality are major, overarching problems in war-related PTSD research. There are scientifically tested strategies from non-military settings and for other mental disorders to improve access to and quality of care; unfortunately, these strategies are unstudied in the military health system and for PTSD and depression. These strategies include care manager coordination (connecting patient, provider, and specialist), collaborative care (negotiated patient-provider problem definition, monitoring of status and treatment response, self-management support, telehealth sustained follow-up), and stepped care (logical, patient-centered and guideline-concordant treatment sequencing). This study aims to fill these gaps and evaluate these systems-level strategies in a military setting for PTSD and depression.

The purpose of the STEPS UP (STepped Enhancement of PTSD Services Using Primary Care) trial is to compare centralized telephonic care management with preference-based stepped PTSD and depression care to optimized usual care. We hypothesize that the STEPS UP intervention will lead to improvements in (1) PTSD and depression symptom severity (primary hypothesis); (2) somatic symptom severity, alcohol use, mental health functioning, work functioning; (3) costs and cost-effectiveness. We further hypothesize that qualitative data obtained from interviews will show that (4) patients, their family members, and participating clinicians find the STEPS-UP intervention to be an acceptable, effective, and satisfying approach to deliver and receive PTSD and depression care.

STEPS-UP is a six-site, two-parallel arm (N = 666) randomized controlled effectiveness trial with 3-month, 6-month, and 12-month follow-up comparing centralized telephonic stepped-care management to optimized usual PTSD and depression care. In addition to the existing PTSD and depression treatment options, STEPS UP includes web-based cognitive behavioral self-management, telephone cognitive-behavioral therapy, continuous RN nurse care management, and computer-automated care management support. Both arms can refer patients for mental health specialty care as needed, preferred and available. The study uses sites currently running RESPECT-Mil, the existing military primary care-mental health services practice network, to access site health care leaders and potential study participants at the 6 study sites.

If effective, we expect that STEPS UP will increase the percentage of military personnel with unmet PTSD- and depression-related health care needs who get timely, effective, and efficient PTSD and depression care. Our real-world primary care effectiveness emphasis will prevent the Institute of Medicine's so called "15 year science to service gap." If successful, STEPS UP could roll out immediately, reinforcing and facilitating pathways to PTSD and depression recovery.

ELIGIBILITY:
Inclusion Criteria:

* Active duty status at the time of enrollment
* Positive PTSD screen (2 or more yes responses on PC-PTSD), per routine primary care screening.
* DSM-IV-TR criteria for A) PTSD using the PCL-C (i.e.., a "moderate" or greater severity level on 1 re-experiencing, 3 avoidance, and 2 hyperarousal symptoms) and/or B) Depression, using the PHQ-9 (i.e., endorsement of at least 5 of the 9 symptoms experienced "more than half the days" and at least one of those symptoms must include either "little interest or pleasure in doing things" or "feeling down, depressed or hopeless")
* Report of routine computer, Internet, and e-mail access
* Capacity to consent to participation and provide research informed consent using local IRB-approved form

Exclusion Criteria:

* Treatment refractory PTSD or depression after participation in RESPECT-mil or specialty mental health treatment.
* Acute psychosis, psychotic episode, or psychotic disorder diagnosis by history within the past 2 years
* Bipolar I disorder by history or medical record review within last 2 years.
* Active substance dependence disorder in the past year by history within the past 12 months.
* Active suicidal ideation within the past 2 months by history.
* Patients on psychoactive medication, unless that medication dosing and administration has been stable and regular for at least 1 month.
* Acute or unstable physical illness.
* Anticipated deployment, demobilization, or separation during the next six months.
* Personnel who work in participating clinics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Diagnostic Scale (PDS) | baseline - 3 months
  The PDS (Foa, 1996) is a 49-item self-report measure that assesses both severity of PTSD symptoms related to a single identified traumatic event and probable diagnosis of PTSD.
Posttraumatic Diagnostic Scale (PDS) | baseline - 6 months
  The PDS (Foa, 1996) is a 49-item self-report measure that assesses both severity of PTSD symptoms related to a single identified traumatic event and probable diagnosis of PTSD.
Posttraumatic Diagnostic Scale (PDS) | baseline - 12 months
  The PDS (Foa, 1996) is a 49-item self-report measure that assesses both severity of PTSD symptoms related to a single identified traumatic event and probable diagnosis of PTSD.
Hopkins Symptom Checklist Depression Scale-20 Item Version (HSCL-20) | baseline - 3 months
  The HSCL-20 is a self-report scale comprising the 13 items of the Hopkins Symptom Checklist Depression Scale plus 7 additional items from the Hopkins Symptom Checklist-90-Revised. The HSCL-20 has been widely used as an outcome measure of depressive severity in large clinical trials (Boudreau, et al., 2002; Felker, et al., 2001; Fraser, et al., 2004; Hedrick, et al., 2003; Katon, et al., 1996; Kroenke, et al., 2001; Unutzer, et al., 2002; Williams, et al., 2000).
Hopkins Symptom Checklist Depression Scale-20 Item Version (HSCL-20) | baseline - 6 months
  The HSCL-20 is a self-report scale comprising the 13 items of the Hopkins Symptom Checklist Depression Scale plus 7 additional items from the Hopkins Symptom Checklist-90-Revised. The HSCL-20 has been widely used as an outcome measure of depressive severity in large clinical trials (Boudreau, et al., 2002; Felker, et al., 2001; Fraser, et al., 2004; Hedrick, et al., 2003; Katon, et al., 1996; Kroenke, et al., 2001; Unutzer, et al., 2002; Williams, et al., 2000).
Hopkins Symptom Checklist Depression Scale-20 Item Version (HSCL-20) | baseline - 12 months
  The HSCL-20 is a self-report scale comprising the 13 items of the Hopkins Symptom Checklist Depression Scale plus 7 additional items from the Hopkins Symptom Checklist-90-Revised. The HSCL-20 has been widely used as an outcome measure of depressive severity in large clinical trials (Boudreau, et al., 2002; Felker, et al., 2001; Fraser, et al., 2004; Hedrick, et al., 2003; Katon, et al., 1996; Kroenke, et al., 2001; Unutzer, et al., 2002; Williams, et al., 2000).

SECONDARY OUTCOMES:
Somatic Symptom Severity - Patient Health Questionnaire - 15 (PHQ-15) | baseline - 3 months
  Somatic symptom severity will be measured with the widely used and validated 15 item Patient Health Questionnaire (PHQ-15; Kroenke, Spitzer, & Williams, 2002). A total sum of greater than or equal to 15 indicate a high somatic symptom severity based on data from primary care settings (Kroenke et al., 2002).
Somatic Symptom Severity - Patient Health Questionnaire - 15 (PHQ-15) | baseline - 6 months
  Somatic symptom severity will be measured with the widely used and validated 15 item Patient Health Questionnaire (PHQ-15; Kroenke, Spitzer, & Williams, 2002). A total sum of greater than or equal to 15 indicate a high somatic symptom severity based on data from primary care settings (Kroenke et al., 2002).
Somatic Symptom Severity - Patient Health Questionnaire - 15 (PHQ-15) | baseline - 12 months
  Somatic symptom severity will be measured with the widely used and validated 15 item Patient Health Questionnaire (PHQ-15; Kroenke, Spitzer, & Williams, 2002). A total sum of greater than or equal to 15 indicate a high somatic symptom severity based on data from primary care settings (Kroenke et al., 2002).
Alcohol Use Disorders Identification Test (AUDIT) | eligibility - 3 months
  The AUDIT (Babor, Higgins-Biddle, Saunders, & Monteiro, 2001) will be used to assess alcohol use, alcohol dependence symptoms, and alcohol-related problems, focused on the recent past. This 10-item scale is widely used and has been shown to be consistent with ICD-10 definitions for alcohol dependence and harmful alcohol use (Allen, Litten, Fertig, & Babor, 1997; Saunders, Aasland, Amundsen, & Grant, 1993; Saunders, Aasland, Babor, de, & Grant, 1993)
Alcohol Use Disorders Identification Test (AUDIT) | eligibility - 6 months
  The AUDIT (Babor, Higgins-Biddle, Saunders, & Monteiro, 2001) will be used to assess alcohol use, alcohol dependence symptoms, and alcohol-related problems, focused on the recent past. This 10-item scale is widely used and has been shown to be consistent with ICD-10 definitions for alcohol dependence and harmful alcohol use (Allen, Litten, Fertig, & Babor, 1997; Saunders, Aasland, Amundsen, & Grant, 1993; Saunders, Aasland, Babor, de, & Grant, 1993)
Alcohol Use Disorders Identification Test (AUDIT) | eligibility - 12 months
  The AUDIT (Babor, Higgins-Biddle, Saunders, & Monteiro, 2001) will be used to assess alcohol use, alcohol dependence symptoms, and alcohol-related problems, focused on the recent past. This 10-item scale is widely used and has been shown to be consistent with ICD-10 definitions for alcohol dependence and harmful alcohol use (Allen, Litten, Fertig, & Babor, 1997; Saunders, Aasland, Amundsen, & Grant, 1993; Saunders, Aasland, Babor, de, & Grant, 1993)
Health-Related Quality of Life and Functional Status - Medical Outcomes Study Short Form-12 (SF-12) | baseline - 3 months
  Limitations in role functioning will be assessed using the SF-12 (Ware et al., 1996). The SF-12 is a widely used measure of health-related quality of life and functioning with established reliability and validity. This measure will be used for the economic analysis as well as to measure functioning as an outcome.
Health-Related Quality of Life and Functional Status - Medical Outcomes Study Short Form-12 (SF-12) | baseline - 6 months
  Limitations in role functioning will be assessed using the SF-12 (Ware et al., 1996). The SF-12 is a widely used measure of health-related quality of life and functioning with established reliability and validity. This measure will be used for the economic analysis as well as to measure functioning as an outcome.
Health-Related Quality of Life and Functional Status - Medical Outcomes Study Short Form-12 (SF-12) | baseline - 12 months
  Limitations in role functioning will be assessed using the SF-12 (Ware et al., 1996). The SF-12 is a widely used measure of health-related quality of life and functioning with established reliability and validity. This measure will be used for the economic analysis as well as to measure functioning as an outcome.
WHO Health and Work Performance Questionnaire-Short Form (HPQ-SF) | baseline - 3 months
  The HPQ-SF (Kessler, et al., 2004; Kessler, et al., 2003) will be used to assess work presenteeism and absenteeism. The self-report survey contains 11 items and assesses work in the prior 4 weeks. These items will be used both to assess work functioning and to estimate costs related to PTSD and associated conditions.
WHO Health and Work Performance Questionnaire-Short Form (HPQ-SF) | baseline - 6 months
  The HPQ-SF (Kessler, et al., 2004; Kessler, et al., 2003) will be used to assess work presenteeism and absenteeism. The self-report survey contains 11 items and assesses work in the prior 4 weeks. These items will be used both to assess work functioning and to estimate costs related to PTSD and associated conditions.
WHO Health and Work Performance Questionnaire-Short Form (HPQ-SF) | baseline - 12 months
  The HPQ-SF (Kessler, et al., 2004; Kessler, et al., 2003) will be used to assess work presenteeism and absenteeism. The self-report survey contains 11 items and assesses work in the prior 4 weeks. These items will be used both to assess work functioning and to estimate costs related to PTSD and associated conditions.
Numeric Rating Scale for Pain | baseline - 3 months
  This trial will use a two-item numeric rating scale for pain, adapted from the NRS (Cleeland and Ryan, 1994) and the University of Washington's IMPACT studies. The items ask patients to rate pain intensity on average and how much the pain interferes with their daily activities on 11-point numeric rating scales.
Numeric Rating Scale for Pain | baseline - 6 months
  This trial will use a two-item numeric rating scale for pain, adapted from the NRS (Cleeland and Ryan, 1994) and the University of Washington's IMPACT studies. The items ask patients to rate pain intensity on average and how much the pain interferes with their daily activities on 11-point numeric rating scales.
Numeric Rating Scale for Pain | baseline - 12 months
  This trial will use a two-item numeric rating scale for pain, adapted from the NRS (Cleeland and Ryan, 1994) and the University of Washington's IMPACT studies. The items ask patients to rate pain intensity on average and how much the pain interferes with their daily activities on 11-point numeric rating scales.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Bray, PhD, Principal Investigator — RTI International; Lisa Jaycox, PhD, Principal Investigator — RAND; Bradley E Belsher, PhD, Principal Investigator — United States Department of Defense
Locations (6):
- United States (6):
  - Evans Army Community Hospital, Fort Carson, Colorado
  - Winn Army Community Hospital, Fort Stewart, Georgia
  - Blanchfield Army Community Hospital, Fort Campbell, Kentucky
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - William Beaumont Army Medical Center, Fort Bliss, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engel CC. Improving primary care for military personnel and veterans with posttraumatic stress disorder--the road ahead. Gen Hosp Psychiatry. 2005 May-Jun;27(3):158-60. doi: 10.1016/j.genhosppsych.2005.01.001. No abstract available. PMID 15882761
- [Background] Engel CC, Hyams KC, Scott K. Managing future Gulf War Syndromes: international lessons and new models of care. Philos Trans R Soc Lond B Biol Sci. 2006 Apr 29;361(1468):707-20. doi: 10.1098/rstb.2006.1829. PMID 16687273
- [Background] Spira, J.L., Pyne, J.M., & Wiederhold, B. (2006). Chapter 10: Experiential Methods in the Treatment of Combat PTSD. In Figley, C.R. and Nash, W.P. In For Those Who Bore the Battle: Combat Stress Injury Theory, Research, and Management. For the Routledge Psychosocial Stress Book Series
- [Background] Tanielian, T. & Jaycox, L., Eds. "Invisible Wounds of War: Psychological and Cognitive Injuries, Their Consequences, and Services to Assist Recovery." RAND/MG-720- CCF (available at http://veterans.rand.org)
- [Background] Jaycox LH, Stein BD, Kataoka SH, Wong M, Fink A, Escudero P, Zaragoza C. Violence exposure, posttraumatic stress disorder, and depressive symptoms among recent immigrant schoolchildren. J Am Acad Child Adolesc Psychiatry. 2002 Sep;41(9):1104-10. doi: 10.1097/00004583-200209000-00011. PMID 12218432
- [Background] Lisa S. Meredith, Terri L. Tanielian, Michael D. Greenberg, Ana Suárez, Elizabeth Eiseman. "Expanding Access to Mental Health Counselors: Evaluation of the Tricare Demonstration" RAND/DRR-3458-1-OSD (available at www.rand.org)
- [Background] Stein BD, Tanielian TL, Ryan GW, Rhodes HJ, Young SD, Blanchard JC. A bitter pill to swallow: nonadherence with prophylactic antibiotics during the anthrax attacks and the role of private physicians. Biosecur Bioterror. 2004;2(3):175-85. doi: 10.1089/bsp.2004.2.175. PMID 15588055
- [Background] Meredith LS, Mendel P, Pearson M, Wu SY, Joyce G, Straus JB, Ryan G, Keeler E, Unutzer J. Implementation and maintenance of quality improvement for treating depression in primary care. Psychiatr Serv. 2006 Jan;57(1):48-55. doi: 10.1176/appi.ps.57.1.48. PMID 16399962
- [Background] Litz BT, Engel CC, Bryant RA, Papa A. A randomized, controlled proof-of-concept trial of an Internet-based, therapist-assisted self-management treatment for posttraumatic stress disorder. Am J Psychiatry. 2007 Nov;164(11):1676-83. doi: 10.1176/appi.ajp.2007.06122057. PMID 17974932
- [Background] Williams JW Jr, Gerrity M, Holsinger T, Dobscha S, Gaynes B, Dietrich A. Systematic review of multifaceted interventions to improve depression care. Gen Hosp Psychiatry. 2007 Mar-Apr;29(2):91-116. doi: 10.1016/j.genhosppsych.2006.12.003. PMID 17336659
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Hoge CW, Auchterlonie JL, Milliken CS. Mental health problems, use of mental health services, and attrition from military service after returning from deployment to Iraq or Afghanistan. JAMA. 2006 Mar 1;295(9):1023-32. doi: 10.1001/jama.295.9.1023. PMID 16507803
- [Background] Engel CC, Oxman T, Yamamoto C, Gould D, Barry S, Stewart P, Kroenke K, Williams JW Jr, Dietrich AJ. RESPECT-Mil: feasibility of a systems-level collaborative care approach to depression and post-traumatic stress disorder in military primary care. Mil Med. 2008 Oct;173(10):935-40. doi: 10.7205/milmed.173.10.935. PMID 19160608
- [Result] Engel CC, Bray RM, Jaycox LH, Freed MC, Zatzick D, Lane ME, Brambilla D, Rae Olmsted K, Vandermaas-Peeler R, Litz B, Tanielian T, Belsher BE, Evatt DP, Novak LA, Unutzer J, Katon WJ. Implementing collaborative primary care for depression and posttraumatic stress disorder: design and sample for a randomized trial in the U.S. military health system. Contemp Clin Trials. 2014 Nov;39(2):310-9. doi: 10.1016/j.cct.2014.10.002. Epub 2014 Oct 12. PMID 25311446
- [Result] Belsher BE, Jaycox LH, Freed MC, Evatt DP, Liu X, Novak LA, Zatzick D, Bray RM, Engel CC. Mental Health Utilization Patterns During a Stepped, Collaborative Care Effectiveness Trial for PTSD and Depression in the Military Health System. Med Care. 2016 Jul;54(7):706-13. doi: 10.1097/MLR.0000000000000545. PMID 27111751
- [Result] Engel CC, Jaycox LH, Freed MC, Bray RM, Brambilla D, Zatzick D, Litz B, Tanielian T, Novak LA, Lane ME, Belsher BE, Olmsted KL, Evatt DP, Vandermaas-Peeler R, Unutzer J, Katon WJ. Centrally Assisted Collaborative Telecare for Posttraumatic Stress Disorder and Depression Among Military Personnel Attending Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):948-56. doi: 10.1001/jamainternmed.2016.2402. PMID 27294447
- [Result] Tanielian T, Woldetsadik MA, Jaycox LH, Batka C, Moen S, Farmer C, Engel CC. Barriers to Engaging Service Members in Mental Health Care Within the U.S. Military Health System. Psychiatr Serv. 2016 Jul 1;67(7):718-27. doi: 10.1176/appi.ps.201500237. Epub 2016 Mar 15. PMID 26975521
- [Result] Batka C, Tanielian T, Woldetsadik MA, Farmer C, Jaycox LH. Stakeholder Experiences in a Stepped Collaborative Care Study Within U.S. Army Clinics. Psychosomatics. 2016 Nov-Dec;57(6):586-597. doi: 10.1016/j.psym.2016.05.008. Epub 2016 May 31. PMID 27478057
- [Result] Bray RM, Engel CC, Williams J, Jaycox LH, Lane ME, Morgan JK, Unutzer J. Posttraumatic Stress Disorder in U.S. Military Primary Care: Trajectories and Predictors of One-Year Prognosis. J Trauma Stress. 2016 Aug;29(4):340-8. doi: 10.1002/jts.22119. Epub 2016 Jul 22. PMID 27447948
- [Derived] Belsher BE, Evatt DP, Liu X, Freed MC, Engel CC, Beech EH, Jaycox LH. Collaborative Care for Depression and Posttraumatic Stress Disorder: Evaluation of Collaborative Care Fidelity on Symptom Trajectories and Outcomes. J Gen Intern Med. 2018 Jul;33(7):1124-1130. doi: 10.1007/s11606-018-4451-5. Epub 2018 Apr 27. PMID 29704183